CLINICAL TRIAL: NCT05749263
Title: Sleep Patterns as Predictive Markers of Hospitalization or Death Due to Cardiovascular Disease in Elderly Patients
Brief Title: A Study of Sleep Patterns to Determine Predictive Markers Due to Cardiovascular Disease in Elderly Patients
Status: Terminated | Type: Observational
Why Stopped: Difficulty managing the study from a different state
Sponsor: Mayo Clinic (Other)
Collaborators: Sleep Number Corporation (Unknown)
Responsible Party: Principal Investigator, Amir Lerman, Principal Investigator, Mayo Clinic
Other Study IDs: 22-001110
Record Dates: First submitted 2023-02-16; First posted 2023-03-01 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases
Keywords: Elderly Patients; Sleep Patterns
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to learn if there are predictive markers of hospitalization or death that can be found from data gathered from a Sleep Number® bed. This is a prospective observational cohort study that will follow participating subjects in the Masonic Homes/Acacia Creek Retirement Community in Union City, California.

ELIGIBILITY:
Inclusion Criteria:

* Subjects living at Masonic Homes/Acacia Creek Retirement Community who use a Sleep Number® bed and are cognitively able to consent on their own accord.

Exclusion Criteria:

* Subjects who do not have a Sleep Number® bed.
* Subjects without an internet connection to transmit nightly SleepIQ® data.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants eligible for this study will be people who are living in the Masonic Homes/Acacia Creek Retirement Community in Union City, California and who have Sleep Number® beds that record their nightly sleep and physiologic patterns.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 5 years
  Total number of subject deaths due to medical conditions including congestive heart failure, myocardial infarction, atrial fibrillation and sudden cardiac death.
Number of subject hospitalizations | 5 years
  Total number of subjects that required hospitalization due to medical conditions including congestive heart failure, myocardial infarction, atrial fibrillation, and sudden cardiac death.

SECONDARY OUTCOMES:
Change in daytime sleepiness | Baseline, every 6 months for 5 years
  Measured by Epworth Sleepiness Scale. The test is a list of eight situations in which you rate your tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing. Total score is graded from 0-24. 0-7:It is unlikely that you are abnormally sleepy. 8-9:You have an average amount of daytime sleepiness. 10-15:You may be excessively sleepy depending on the situation. You may want to consider seeking medical attention. 16-24:You are excessively sleepy and should consider seeking medical attention.
Change in alertness | Baseline, every 6 months for 5 years
  Measured by alertness rating scale which ranges from 1-6 with lower scores indicating worse subject alertness and function.
Change in depression symptom severity | Baseline, every 6 months for 5 years
  Measured by the Patient Health Questionnaire (PHQ-8) an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score ranges from 0-24, with a higher score indicating greater depression symptom severity.
Change in sleep quality | Baseline, every 6 months for 5 years
  Measured by Pittsburgh Sleep Quality Index. Individuals items within the index are rated on a scale from 0-3 with higher scores indicating worse sleep quality.
Change in Attention-deficit/hyperactivity disorder (ADHD) symptom severity | Baseline, every 6 months for 5 years
  Measured by Adult ADHD Self-Report Scale. The ADHD Self-Report Scale consists of 18 items designed to rate ADHD inattention and hyperactivity/impulsivity symptoms. Each item is score from 0 to 4, with a total score ranging from 0 to 72 and higher scores indicating greater symptom severity.
Change in Verbal Memory | Baseline, every 6 months for 5 years
  Subjects are tasked with remembering fifteen words, presented one at a time, in a field that contains a total of thirty words (fifteen distractors). Subjects are tested at the beginning of the battery and again near the end. The verbal memory test measures how well subjects can recognize, remember and retrieve words. Low scores indicate verbal memory impairment.
Change in Visual Memory | Baseline, every 6 months for 5 years
  Subjects are tasked with remembering fifteen geometric figures, presented one at a time, in a field with fifteen distractors. Subjects are tested near the beginning of the battery and again at the end. The visual memory test measures a subject's ability to recognize, remember and retrieve shapes. Low scores indicate visual memory impairment.
Change in Motor Skills | Baseline, every 6 months for 5 years
  Measured by the Finger Tapping Test (FTT). The FTT tests motor speed and fine motor control. In it, subjects participate in three rounds of tapping with each hand; lowering scores indicate motor slowing.
Change in Processing Speed | Baseline, every 6 months for 5 years
  Measured by Symbol Digit Coding which draws upon several cognitive processes simultaneously (such as visual scanning, visual perception, visual memory and motor function). Subjects are presented with a simple grid, with numbers corresponding to a particular symbol. Sequences of symbols are then provided, which the subject must render in numerics. Low scores are indicative of slow processing speed, possibly due to cognitive impairment.
Change in Stroop Task | Baseline, every 6 months for 5 years
  The Stroop Task measures how well subjects adapt to rapidly changing (and increasingly complex) sets of directions. Words for various colors (i.e. RED, GREEN) are presented in various font colors, which may or may not correspond (i.e. the word "RED" may be rendered in red, or in green). Subjects are tasked with responding under various conditions, such as when the word is rendered in the corresponding color, or when the word and the color it is rendered in are mismatched. Prolonged reactions times indicate cognitive slowing/impairment.
Change in Executive Function | Baseline, every 6 months for 5 years
  Measured by the Shifting Attention Test (SAT). The SAT measures executive function; specifically, how well a subject recognizes set shifting (mental flexibility) and abstraction (rules, categories), and manages multiple tasks simultaneously. In addition, subjects have to adjust their responses to randomly changing rule sets. Low scores are most indicative of cognitive impairments.
Change in Vigilance | Baseline, every 6 months for 5 years
  Measured by the Continuous Performance Test (CPT). The CPT measures sustained vigilance and choice reaction time. Two errors may be clinically significant, more than four errors is clinically significant and likely indicates attentional dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Masonic Homes of California-Acacia Creek, Union City, California
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials